CLINICAL TRIAL: NCT03112252
Title: App-basierte Patientenbefragung Von Allergiepatienten Unter Medikation in Der Pollenflug-Saison Zur Bestimmung Der Auswirkung Einer Allergischen Rhinitis Auf Die Lebensqualität
Brief Title: App Based Study on the Symptoms of Patients With Allergic Rhinitis in the Pollen Season
Status: Completed | Type: Observational
Sponsor: University Hospital of Cologne (Other)
Responsible Party: Principal Investigator, Prof. Dr. Ralph Mösges, Prof. Dr., University Hospital of Cologne
Other Study IDs: IITMACVIA2017D
Record Dates: First submitted 2017-03-30; First posted 2017-04-13 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Allergic Rhinitis
Keywords: Immunotherapy
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no specifications. Depending on the patients — patients with allergic rhinitis

SUMMARY:
App-based study of allergy patients under medication in the pollen season to determine the effect of allergic rhinitis on the quality of life.

DETAILED DESCRIPTION:
The project aims to determine the effects of rhinitis on everyday life and thereby identify the affected pathways, irrespective of age, gender or gender socioeconomic status to lead a healthy and active life.

ELIGIBILITY:
inclusion criteria patients with allergic rhinitis

exclusion criteria none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with allergic rhinitis
Sampling Method: Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
allergic symptoms of patients | one month
  allergic symptoms of patients during the pollen season

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Mösges, Prof. Dr., Principal Investigator — University Hospital of Cologne
Locations (1):
- Institute of Medical Statistics, Informatics and Epidemiology, Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No